CLINICAL TRIAL: NCT00061334
Title: Social Knowledge Representation in the Human Prefrontal Cortex
Brief Title: Investigating the Cognitive Processes That Underlie Social Knowledge and Behavior
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030196; 03-N-0196
Record Dates: First submitted 2003-05-23; First posted 2003-05-26 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-12-29

CONDITIONS: Healthy
Keywords: Attitudes; fMRI; Development; Stereotypes; Memory; Healthy Volunteer; HV
MeSH Terms: conditions — Behavior; Stereotypic Movement Disorder

SUMMARY:
The purpose of the protocol is to localize the neural regions and systems mediating the forms of knowledge representations hypothesized by the principal investigator to be stored in the human prefrontal cortex. Utilizing a variety of experimental neuropsychological tasks during functional MRI, we will investigate hypotheses regarding the role of the dorsolateral and ventromedial prefrontal cortex in social cognition and emotional processing. We will ascertain the relationship between so-called cold cognition such as event knowledge and "hot" social cognition such as attitude formation and specific brain regions within the prefrontal cortex. We will also attempt to determine the relationship between non-frontal neural structures involved in emotional expressions, such as amygdala, and those frontal neural structures involved in executive functions that may modulate emotion. The data that we collect in this protocol will be of value in (1) identifying a set of neural regions and distributed networks mediating the forms of knowledge representation stored in the prefrontal cortex and (2) developing functional MRI screening measures for subjects at-risk for developing a neurological disorder. We will also use the data obtained in these studies with healthy adult volunteers to constrain theories of frontal lobe function based on the study of patients with focal or diffuse frontal lobe lesions and to provide convergent evidence for the role of specific frontal cortex sectors in specific cognitive functions.

DETAILED DESCRIPTION:
Objective

The purpose of the protocol is to localize the neural regions and systems mediating the forms of knowledge representations hypothesized by the principal investigator to be stored in the human prefrontal cortex. We suspect that political attitudes can also be viewed as a type of stored knowledge. Religious attitudinal and event knowledge are also expected to be similarly represented and stored. Utilizing a variety of experimental neuropsychological tasks during functional MRI, we will investigate hypotheses regarding the role of the dorsolateral and ventromedial prefrontal cortex in social cognition and emotional processing. We will ascertain the relationship between so-called "cold" cognition such as event knowledge and "hot" social cognition such as attitude formation and specific brain regions within the prefrontal cortex.

Study Population

Normal adult volunteers will participate in experiments dealing with processing of event knowledge, general attitudes, political stereotypes and attitudes, and religious attitudes, using fMRI.

Design

All the experiments will employ within-subject event-related fMRI design to determine whether activations of different cortical areas correspond to different kind of stored knowledge.

Outcome Measures

The data that we collect in this protocol will consist of fMRI activation images corresponding to varying neuropsychological tasks. The will be of value in (1) identifying a set of neural regions and distributed networks mediating the forms of knowledge representation stored in the prefrontal cortex and (2) developing functional MRI screening measures for subjects at-risk for developing a neurological disorder.

ELIGIBILITY:
* INCLUSION CRITERIA:

The healthy normal controls recruited into these studies will be determined by Section staff phone and in-person interviews to be free of psychiatric, neurological, or other medical disorders that would constrain interpretation of their performance during functional neuroimaging studies. In addition, all normal volunteers must undergo a neuroexam performed by the medically responsible investigator, an NINDS physician, once a year before undergoing MRI scanning. The neurological exam will be done in the neurology outpatient clinic.

All subjects will be native English-speakers and right-handed, as measured by the Edinburgh Handedness Inventory, due to the association between language lateralization and handedness.

In addition, all subjects in Study 3 (that addresses political stereotypes) will be American and will be screened for political affiliation using several measures prior to participation in the study.

Political affiliation will be assessed by obtaining (1) self-reported political orientation of the subject on a scale of 1 to 7 (where 1 is extremely liberal and 7 is extremely conservative, Wyer et al., 1991), (2) political party preference of the subject on a scale of 1 to 7 (where 1 is strongly Democratic and 7 is strongly Republican, Wyer et al., 1991), and (3) scores on the Conservatism-Liberalism Scale (Mehrabian, 1996). Subjects rating their orientation and preference (measures 1 and 2) as 3 or lower or 5 or higher and also scoring higher than 20 or lower than -20 (maximum scores are plus or minus 28) on the Conservatism-Liberalism Scale will be included in the study. American citizenship and the political screening is necessary to enable the classification of conditions as stereotype-congruent and - incongruent (as this is determined by their status as 'Democrat' or 'Republican'). Subjects in Study 4 (that addresses political psychological structures) will be screened to be American citizens prior to participating to the study. Party affiliation, political orientation and adjunctive demographical data will be collected at the end of the fMRI scan to be eventually considered as a potential source of variability in the statistical analysis.

EXCLUSION CRITERIA:

Individuals with a neurological or psychiatric history or medical condition that would compromise our interpretation of the fMRI results will be excluded.

Exclusion criteria are: medical contraindications to MRI procedures (e.g. pacemakers, cochlear devices, surgical clips); technical contraindications to MRI procedures (e.g. no braces); CNS active medications; and claustrophobia.

Pregnant women will also be excluded from participation due to the unknown effects of the high magnetic field on a developing fetus; to ensure compliance with this criterion, all women will undergo a pregnancy test within 24 hours prior to the scan. The results of the pregnancy test must be negative in order for the women to be scanned.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2003-05-07; Study Completion 2011-12-29

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Cordes D, Turski PA, Sorenson JA. Compensation of susceptibility-induced signal loss in echo-planar imaging for functional applications. Magn Reson Imaging. 2000 Nov;18(9):1055-68. doi: 10.1016/s0730-725x(00)00199-5. PMID 11118760
- [Background] Deichmann R, Josephs O, Hutton C, Corfield DR, Turner R. Compensation of susceptibility-induced BOLD sensitivity losses in echo-planar fMRI imaging. Neuroimage. 2002 Jan;15(1):120-35. doi: 10.1006/nimg.2001.0985. PMID 11771980
- [Background] Desmond JE, Glover GH. Estimating sample size in functional MRI (fMRI) neuroimaging studies: statistical power analyses. J Neurosci Methods. 2002 Aug 30;118(2):115-28. doi: 10.1016/s0165-0270(02)00121-8. PMID 12204303